CLINICAL TRIAL: NCT01858714
Title: Environmental and Acceptance-Based Innovations for Weight Loss Maintenance
Acronym: ENACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Meghan Butryn, Ph.D., Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK092374 (NIH)
Record Dates: First submitted 2012-06-19; First posted 2013-05-21 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: obesity; overweight; weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Behavior Therapy; Environment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavior Therapy (BT) (Active Comparator): Active Comparator: Behavior Therapy
  Behavioral treatment strategies will be utilized to facilitate adherence to the treatment goals in all three treatments. Participants in the BT condition will receive only the BT intervention. Strategies that will be emphasized are listed below:
  Self monitoring Stimulus control Changing eating behaviors Goal setting Problem solving Social support Cognitive restructuring Relapse prevention
  Interventions: Behavioral: Behavior Therapy for Weight Loss
- Behavior Therapy + Environment (Experimental): Participants will receive standard behavioral therapy with an emphasis on environmental strategies.
  Interventions: Behavioral: Behavior Therapy + Environment
- Acceptance-based BT + Environment (Experimental): Participants will receive acceptance-based behavioral therapy with an emphasis on environmental strategies.
  Interventions: Behavioral: Acceptance-based Behavior Therapy + Environment

INTERVENTIONS:
Behavioral: Behavior Therapy for Weight Loss — Standard behavioral treatment for weight loss and weight loss maintenance.
  Arms: Behavior Therapy (BT)
Behavioral: Behavior Therapy + Environment — Standard behavioral therapy with an emphasis on environmental strategies.
  Arms: Behavior Therapy + Environment
Behavioral: Acceptance-based Behavior Therapy + Environment — Behavioral therapy with acceptance-based and environmental strategies.
  Arms: Acceptance-based BT + Environment

SUMMARY:
The major goal of this project is to evaluate an innovative approach to obesity involving modification of the home environment. The project also will evaluate if home environment modification is more effective when supplemented with distress tolerance and related skills training.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI between 27 and 45 kg/m2
* Have the ability to engage in physical activity (i.e., can walk at least 2 blocks without stopping for rest)
* Successfully complete all steps in the enrollment process, including completion of a 7-day food diary and attendance at all pre-randomization clinic visits

Exclusion Criteria:

* Have a medical condition (e.g., cancer) or psychiatric condition (e.g., psychotic disorder, substance dependence, bulimia nervosa) that may limit their ability to comply with the behavioral recommendations of the program or pose a risk to the participant during weight loss
* Are pregnant or plan to become pregnant in next 2 years
* Report recently beginning a course of or changing the dosage of prescription medications that can cause significant weight loss or weight gain
* Are participating in or plan to participate in another weight loss program in the next 2 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2011-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, 6 months, 12 months, 18 months, 24 months
Change in Physical Activity | Baseline, 6 months, 12 months, 18 months, 24 months
  Objectively measured physical activity will be recorded at each time point.
Change in Nutritional Intake | Baseline, 12 months, 24 months
  Measured by 24-hour food recall
Change in Psychosocial Status | Baseline, 6 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chabria R, Hagerman CJ, Crane N, Ehmann M, Knudsen FM, Brown KL, Forman E, Butryn ML. Racial disparities in the efficacy of traditional versus acceptance-based behavioral weight loss. Health Psychol. 2025 Jul 24:10.1037/hea0001537. doi: 10.1037/hea0001537. Online ahead of print. PMID 40705619
- [Derived] Butryn ML, Call CC, Schumacher LM, Kerrigan SG, Forman EM. Time to Peak Weight Loss During Extended Behavioral Treatment. Obesity (Silver Spring). 2018 Apr;26(4):658-664. doi: 10.1002/oby.22127. Epub 2018 Feb 14. PMID 29442440
- [Derived] Butryn ML, Forman EM, Lowe MR, Gorin AA, Zhang F, Schaumberg K. Efficacy of environmental and acceptance-based enhancements to behavioral weight loss treatment: The ENACT trial. Obesity (Silver Spring). 2017 May;25(5):866-872. doi: 10.1002/oby.21813. Epub 2017 Mar 23. PMID 28337847
- [Derived] Butryn ML, Arigo D, Raggio GA, Kaufman AI, Kerrigan SG, Forman EM. Measuring the Ability to Tolerate Activity-Related Discomfort: Initial Validation of the Physical Activity Acceptance Questionnaire (PAAQ). J Phys Act Health. 2015 May;12(5):717-6. doi: 10.1123/jpah.2013-0338. Epub 2014 Aug 7. PMID 25106049